CLINICAL TRIAL: NCT04449198
Title: Type 1 Diabetes, Endothelin, and Skeletal Muscle Mitochondrial Dysfunction: The Role of Sirtuin-1
Acronym: T-St1M
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Ryan Harris, Associate Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1595933
Record Dates: First submitted 2020-06-11; First posted 2020-06-26 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; heart disease; muscle function; blood vessels
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Heart Diseases | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Individuals with type 1 diabetes (Experimental): Individuals with type 1 diabetes will be randomly assigned to 1 of the 2 interventions (Resveratrol or placebo)
  Interventions: Drug: Resveratrol; Other: Placebo
- Healthy Controls (No Intervention): Healthy individuals who participate will receive no intervention and serve as controls.

INTERVENTIONS:
Drug: Resveratrol — 500 mg of oral trans-resveratrol twice daily (in the morning and evening) for 12-weeks
  Arms: Individuals with type 1 diabetes
Other: Placebo — placebo for 12 weeks
  Arms: Individuals with type 1 diabetes

SUMMARY:
The proposed study is designed to test the hypothesis that treatment of resveratrol for 12 weeks will improve both endothelin-B receptor (aim 1) and skeletal muscle mitochondrial function (aim 2) in people with type 1 diabetes.

DETAILED DESCRIPTION:
Preliminary data from the investigators' laboratory demonstrate a negative relationship between hemoglobin A1c (HbA1c) and ETBR function, supporting ETBR may be dysfunctional in the presence of T1D. Using near infrared spectroscopy (NIRS) to non-invasively assess muscle function, the investigators have also observed reduced skeletal muscle mitochondrial function in people with T1D compared to healthy controls. In addition, reduced circulating Sirt1 is associated with both ETBR and skeletal muscle mitochondrial dysfunction in the general population. For the current application, the investigators propose to utilize intradermal microdialysis and NIRS as unique, novel, and minimally invasive methods to investigate ETBR and skeletal muscle mitochondrial function, respectively, in people with T1D. Accordingly, the central hypothesis is that increasing circulating Sirt1 with oral supplementation of resveratrol will improve both ETBR function and mitochondrial skeletal muscle function, reducing overall CVD risk (Figure 1). The investigators will test this hypothesis with the following specific aims:

Aim 1: To test the hypothesis that an increase in Sirt1 will improve ETBR function in people with T1D. The investigators will evaluate ETBR function and circulating Sirt1 at baseline and after a 12-week treatment of resveratrol or placebo. Based on preliminary data, the investigators predict that people with T1D will have ETBR dysfunction compared to controls. In addition, the investigators predict that increasing Sirt1 following resveratrol treatment will improve ETBR function, whereas no change will occur with placebo.

Aim 2: To test the hypothesis that an increase in Sirt1 will improve skeletal muscle mitochondrial function and lower HbA1c in people with T1D. A non-invasive assessment of skeletal muscle function will be performed on people with T1D before and after 12-weeks of treatment with resveratrol or placebo. Compared to controls, the investigators predict that people with T1D will have skeletal muscle dysfunction. Following 12 weeks of resveratrol, the investigators predict that the increase in circulating Sirt1 will improve skeletal muscle function. Additionally, the investigators predict the improved skeletal muscle function will contribute to a subsequent decrease in HbA1c in people with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Men and premenopausal women
* All races
* Clinical diagnosis of insulin-dependent type 1 diabetes (patients only)

Exclusion Criteria:

* Clinical diagnosis of hepatic, cardiovascular, or renal disease
* Uncontrolled diabetes (HbA1C >12%)
* Diabetic complications (i.e. neuropathy)
* Uncontrolled hypertension (>140/90 mm Hg on therapy)
* Pregnancy
* Use of vasoactive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in AUC for ET-1 + BQ-123 | Measure taken at Baseline and post 12 weeks
  Change in Area Under the Curve (AUC) for Cutaneous Vascular Conductance (CVC) in response to co-perfusion of ET-1 + BQ-123 at 12 weeks. Measured using intradermal microdialysis technique in conjunction with Laser Speckle Contrast Imaging (Moor FLPI-2) and beat-by-beat blood pressure monitoring (Finapres NOVA).
Skeletal Muscle Mitochondrial Function | Measure taken at Baseline and post 12 weeks
  Change in Skeletal Muscle Mitochondrial Function at 12 weeks. Measured using Near Infrared Spectroscopy (NIRS). Values are an index of phosphocreatine recovery expressed as a rate constant (min-1)

SECONDARY OUTCOMES:
Change in Percentage Flow-Mediated Dilation (FMD) | Measure taken at Baseline and post 12 weeks
  Change in Percentage FMD at 12 weeks. Measured via ultrasound in conjunction with edge detection software. Expressed as %
Change in Pulse Wave Velocity (PWV) | Measure taken at Baseline and post 12 weeks
  Change in PWV at 12 weeks. Measured by Shygmocor Xcel in m/s.
Change in Post Occlusive Reactive Hyperemia (PORH) | Baseline and post 12 weeks
  Change in PORH at 12 weeks. Measured by Laser Speckle Contrast Imager (Moor FLPI-2) in perfusion units (PU). Represents the maximal dilatory response in the microcirculation post 5 minute occlusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University/Georgia Prevention Institute/ Laboratory of Integrative and Exercise Physiology, Augusta, Georgia, United States

REFERENCES:
- [Derived] Derella CC, Thomas J, Harris RA. Women Have Greater Endothelin-B Receptor Function and Lower Mitochondrial Capacity Compared to Men With Type 1 Diabetes. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2561-2568. doi: 10.1210/clinem/dgad189. PMID 37009678